CLINICAL TRIAL: NCT02630134
Title: MyHealthTrendsTM Device for Pain for Monitoring Pain During the Intraoperative, Pre and Post Surgical Periods: Comparison With Standard of Care Pain Monitoring.
Brief Title: Device for Monitoring Pain During Intraoperative, Pre/Post Surgical Periods: Comparison With Standard of Care Monitoring
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped, recruitment difficult, subject compliance very difficult.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 11-00520
Record Dates: First submitted 2014-04-02; First posted 2015-12-15 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Pain Measurement; Assessment, Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Baeta (Experimental): These patients receive the Baeta device and take it home.
  Interventions: Other: These patients receive the Baeta device and take it home

INTERVENTIONS:
Other: These patients receive the Baeta device and take it home

SUMMARY:
Study patients are given a hand held device to track pain post surgery.

DETAILED DESCRIPTION:
The MyHealthTrends™ for Pain Tracking System is a revolutionary consumer-oriented pain monitoring system enabling individuals to record the pain participants experience with the click of a button. Developed by a doctor for the ultimate use within hospital and outpatient settings, MyHealthTrends™ for Pain enables anyone afflicted with pain to easily record their sensations - helping to acquire faster and superior diagnoses and treatment. Among the benefits of the MyHealthTrends™ for Pain Tracking System are that it enables patients to: i] easily record the pain experienced in real-time - capturing accurate information; ii] shift from memory-based descriptions of experienced pain to data-driven, time based recordings; iii] provide objective evidence of the pain experienced.

It is extremely portable and convenient to carry, approximately the size of a modern automobile key. Since it can be uploaded to a confidential internet site by way of a computer, which site is then accessible to the physician, it provides various additional benefits. These include allowing the physician to: i] identify breakthrough pain episodes; ii] determine analgesic requirements with a real time detailed pain record; iii] prescribe the appropriate regimen with confidence; and iv] monitor pain levels experienced by the patient, free of distortion caused by memory biases and lapses.

The purpose of this study is to provide detailed and quantitative comparisons of the device's performance during a demanding clinical inpatient surgery episode, where standard pain monitoring and therapy are in use. The device is extremely easy to use involving merely the press of a button; and so it would not distract from any standard communication of pain symptoms, which the subject were inclined to convey. The device stores all information (time and date stamped) for downloading through a USB plug to a computer when the study is completed and the patient discharged.

Specifically, investigators will identify 40 post thoracotomy patients expected to receive a PCA or epidural for post op pain control at Tisch hospital. Patients will be given the device and asked to record their pain in the immediate post op period until discharge. The information obtained from the electronic diary will be correlated with pain records based on nurse's chart, administration of pain medication, VAS pain questionnaire instruments given daily to each patient, and call button utilization.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* post thoracotomy with a consult placed to the acute pain service on post-op day 0 for management of a PCA or epidural
* mental status permits patient to reliably press a button to record pain or administer medications
* must be hemodynamically stable
* must be able to physically use the MyHealth trends diary (press a button)
* supplies written informed consent.

Exclusion Criteria:

* less than 18 years of age
* has any underlying or current medical condition, which, in the opinion of the Investigator, would interfere with the use of the MyHealth trends device (e.g. severe psychosis, quadrapalegic, etc.)
* Subject necessitates ICU care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Pain score | 13 days
  VAS score 0-10

SECONDARY OUTCOMES:
Compare regression of Baeta Daily Pain scores | 13 days
  Interpatient comparison of regression of Baeta Daily Pain Score as a function of VAS score
  - Correlation of inpatient and outpatient scores with chart indications of pain, VAS scores and observer scoring of pain behavior (none, mild, moderate, severe).
Correlation of inpatient and outpatient scores with chart indications of pain, VAS scores and observer scoring of pain behavior | 13 days
  Comparing the patient's own scores and observers scoring the subject's pain
Number of cases in which the MHTTM for Pain is superior to standard pain monitoring techniques | 13 days
  Patients whose use indicated that the MHT TM is a better indicator of pain than standard techniques
Number of cases in which the MHTTM for Pain is inferior to standard pain monitoring techniques | 13 days
  Patients whose use indicated MHT TM was an inferior indicator of pain than standard techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Haile, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaertner J, Elsner F, Pollmann-Dahmen K, Radbruch L, Sabatowski R. Electronic pain diary: a randomized crossover study. J Pain Symptom Manage. 2004 Sep;28(3):259-67. doi: 10.1016/j.jpainsymman.2003.12.017. PMID 15336338
- [Background] Marceau LD, Link C, Jamison RN, Carolan S. Electronic diaries as a tool to improve pain management: is there any evidence? Pain Med. 2007 Oct;8 Suppl 3:S101-9. doi: 10.1111/j.1526-4637.2007.00374.x. PMID 17877520